CLINICAL TRIAL: NCT03800797
Title: Efficacy and Safety of Loxoprofen Hydrogel Patch Versus Loxoprofen Tablet in Patients With Ankylosing Spondylitis: a 4-week Randomized, Open-label Study
Brief Title: Efficacy and Safety of Loxoprofen Hydrogel Patch in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gu Jieruo, Director, Department of Rheumatology, The Third Affiliated Hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2014]2-135
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2015-12

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; loxoprofen; patch
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — loxoprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LX-P group (Experimental): loxoprofen sodium hydrogel patch (LX-P) 100 mg per day for 4 weeks
  Interventions: Drug: Loxoprofen sodium hydrogel patch
- LX-T group (Active Comparator): loxoprofen sodium tablet (LX-T) 60 mg t.i.d. for 4 weeks
  Interventions: Drug: Loxoprofen sodium tablet

INTERVENTIONS:
Drug: Loxoprofen sodium hydrogel patch — 100 mg per day
  Other Names: Loxoprofen hydrogel patch
  Arms: LX-P group
Drug: Loxoprofen sodium tablet — 60 mg t.i.d.
  Other Names: Loxoprofen tablet
  Arms: LX-T group

SUMMARY:
To assess the efficacy and safety of loxoprofen sodium hydrogel patch (LX-P) versus loxoprofen sodium tablet (LX-T) in patients with active ankylosing spondylitis(AS). The trial includes 70 patients who are randomly assigned to either the LX-P group (LX-P 100 mg per day) or LX-T group (LX-T 60 mg t.i.d.) for 4 weeks.

DETAILED DESCRIPTION:
This is a 4-week randomized, open-label trial to investigate the efficacy and safety of loxoprofen sodium hydrogel patch (LX-P) versus loxoprofen sodium tablet (LX-T) in patients with active ankylosing spondylitis(AS). The trial includes 70 patients who are randomly assigned to either the LX-P group (LX-P 100 mg per day) or LX-T group (LX-T 60 mg t.i.d.) for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years
* Meet 1984 modified New York criteria for AS
* The Bath AS Disease Activity Index (BASDAI) ≥4 on a 0-10-cm visual analog scale or the Ankylosing Spondylitis Disease Activity Score using the C-reactive protein level (ASDAS-CRP) ≥1.3
* NSAIDs washout period of at least 5 days prior to randomization
* DMARDs washout period of at least 4 weeks prior to randomization
* Corticosteroids washout period of at least 4 weeks prior to randomization
* Biological agents washout period of at least 3 months prior to randomization.

Exclusion Criteria:

* Peptic ulcer
* Unstable cardiac diseases
* Abnormal hepatic function with an elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 times of upper normal limits
* Abnormal renal function with creatinine more than upper normal limit
* Hematologic disorders
* Psychosis
* Malignancy
* Allergic to LX drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
the proportions of patients reaching Assessment in Ankylosing Spondylitis 20% response (ASAS20) | week 4
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥1 unit (0-10-cm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (mean of total and nocturnal pain scores), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)

SECONDARY OUTCOMES:
ASAS5/6 response | week 4
  defined as 20% improvement in 5 of the following 6 domains: PTGA, pain assessment, BASFI, clinical inflammation, spinal mobility, and C-reactive protein (CRP)
ASAS20 response | week 2
  ASAS20 was defined as an improvement of ≥20% and absolute improvement of ≥1 unit (0-10-cm VAS) from baseline in ≥3 of the following 4 domains (and absence of deterioration in any domain): patient's global assessment of disease activity (PTGA), pain assessment (mean of total and nocturnal pain scores), Bath Ankylosing Spondylitis Functional Index (BASFI), and clinical inflammation (mean of 2 morning stiffness-related scores on the BASDAI)
ASAS5/6 response | week 2
  defined as 20% improvement in 5 of the following 6 domains: PTGA, pain assessment, BASFI, clinical inflammation, spinal mobility, and C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, Prof, Study Director — Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China